CLINICAL TRIAL: NCT04056273
Title: Assessment of the Use of Radial Endobronchial Ultrasonography With a Guide Sheath in Increasing the Yield Rate of Transbronchial Lung Biopsy
Brief Title: Assess the Use of rEBUS With a Guide Sheath to Increase Transbronchial Lung Biopsy Yield Rate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 201904072RINC
Record Dates: First submitted 2019-08-11; First posted 2019-08-14 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Diagnoses Disease; Lung Tumor
Keywords: guide sheath, bronchoscopic biopsy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guide sheath group (Experimental): Transbronchial biopsy with a guide sheath
  Interventions: Other: Guide sheath group
- Conventional group (Active Comparator): Transbronchial biopsy without a guide sheath
  Interventions: Other: Conventional group

INTERVENTIONS:
Other: Guide sheath group — After the lesion was found by rEBUS, insert the rEBUS into a guide sheath and re-locate the lesion. Fix the guide sheath at that position and perform transbronchial biopsy and brushing through the guide sheath.
  Arms: Guide sheath group
Other: Conventional group — After the lesion was found by rEBUS, mark the location and depth. Insert the biopsy forceps and cytology brush to the marked depth of that bronchiole to perform biopsy and brushing.
  Arms: Conventional group

SUMMARY:
Whether using a guide sheath can increase the diagnostic yield rate after the lesion is located by radial endobronchial ultrasound

DETAILED DESCRIPTION:
For lung nodules, there are several ways to acquire tissue for pathology study, including computed tomography (CT)-guided core needle biopsy, radial probe endobronchial ultrasound (rEBUS)-guided transbronchial lung biopsy (TBLB), convex probe EBUS transbronchial needle aspiration (TBNA), and echo-guided core needle biopsy. rEBUS-guided TBLB has relatively low limitation of lesion position, comparing to echo-guided core needle biopsy and EBUS-TBNA, and doesn't need to deal with the risk of radiation exposure.1 For peripheral pulmonary lesions (PPL), it has good yield rate and the operation is easy.2 However, when bleeding occurs, the procedure time is prolonged for hemostasis. Nonetheless, using a guide sheath can help with the problem. According to the literatures, biopsy yield rates vary but on average it is higher with a guide sheath (62~90% vs. 41~73%), while the complication rates are about the same (1.3~4.4% 1.5~5.0%). The investigators would like to know whether the diagnostic rate is higher with a guide sheath and so do the procedure time and the complication rate. Whether the lesion character affect the yield rate will also be studied.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 20 years old. Radiographic evidence of peripheral pulmonary lesions. The lesion can be located by radial probe EBUS.

Exclusion Criteria:

B1 bronchus. Thrombocytopenia with platelet count < 100K. Coagulopathy with INR > 1.3. High oxygen demand (O2 mask > 28%, 5L). Currently using anti-platelet drug or anti-coagulant.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
The diagnostic yield rate i. Brushing cytology ii. Biopsy | 2 years
  The diagnostic yield rate of transbronchial biopsy and brushing cytology by using guide sheath

SECONDARY OUTCOMES:
Procedure duration | 1 year
  The procedure time of using a guide sheath
Complication rate (pneumothorax, hemoptysis) | 1 year
  The complication rate of using a guide sheath

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chi Ho, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dhooria S, Sehgal IS, Gupta N, Aggarwal AN, Behera D, Agarwal R. Role of radial endobronchial ultrasound-guided transbronchial needle aspiration in the diagnosis of pulmonary nodules: Case report and literature review. Lung India. 2017 Jan-Feb;34(1):61-64. doi: 10.4103/0970-2113.197094. PMID 28144062
- [Result] Eom JS, Mok JH, Kim I, Lee MK, Lee G, Park H, Lee JW, Jeong YJ, Kim WY, Jo EJ, Kim MH, Lee K, Kim KU, Park HK. Radial probe endobronchial ultrasound using a guide sheath for peripheral lung lesions in beginners. BMC Pulm Med. 2018 Aug 13;18(1):137. doi: 10.1186/s12890-018-0704-7. PMID 30103727
- [Result] Hayama M, Okamoto N, Suzuki H, Tamiya M, Shiroyama T, Tanaka A, Nishida T, Nishihara T, Uehara N, Morishita N, Kawahara K, Hirashima T. Radial endobronchial ultrasound with a guide sheath for diagnosis of peripheral cavitary lung lesions: a retrospective study. BMC Pulm Med. 2016 May 11;16(1):76. doi: 10.1186/s12890-016-0244-y. PMID 27170169